CLINICAL TRIAL: NCT06570278
Title: Role of High-Throughput Whole Genome Sequencing for the Diagnosis and Care of Atypical Diabetes
Acronym: GLUCOGEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Commissariat A L'energie Atomique (Other Government); Rennes University Hospital (Other); Central Hospital, Nancy, France (Other); Nantes University Hospital (Other); Imagine Institute (Other); APHP (Other); Hospices Civils de Lyon (Other); Université Lumière Lyon 2 (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C17-27; 2021-A02597-34 (Other: ANSM)
Record Dates: First submitted 2024-02-02; First posted 2024-08-26 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
Keywords: Next generation sequencing genome; Diagnostic study; Medico-economic study
MeSH Terms: conditions — Diabetes Mellitus; Disease

STUDY DESIGN:
Intervention Model Description: We plan to randomize one patient in the control group for two in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control procedure (No Intervention): In-silico analysis of a panel of validated genes (ISApanel). Patients recruited along control procedure will stay in their arm using current genetic diagnosis practices and standard of care that may differ from one center to another
- intervention procedure (Experimental): WGS coupled with MCM
  Interventions: Diagnostic Test: WGS coupled with MCM

INTERVENTIONS:
Diagnostic Test: WGS coupled with MCM — Whole genome will be screened and analysis will focus on pathogenic and likely pathogenic variants. The list of variants of interest will be recorded until examination and discussion during the MCM. MCM will edit a final synthesis concerning the pathogenicity of identified variants.
  Arms: intervention procedure

SUMMARY:
The main objective of the study is to assess the contribution of whole genome sequencing (WGS) coupled with a multidisciplinary conciliation meeting (MCM) on diagnosis of atypical forms of diabetes compared to an in-silico analysis of a panel of validated genes (ISApanel), corresponding to current practice, in a randomized trial.

Notably, the questions it aims to answer are:

* The feasibility of the WGS coupled with MCM on diagnosis of atypical forms of diabetes,
* The contribution of WGS coupled with MCM on number of genetic alterations likely causal of diabetes identified and with a modification in care and support of patients.

After inclusion and sampling for genotyping, patients will be followed for 5 years.

The target population is 1020 adults with atypical diabetes for whom it is possible to obtain a blood sample.

DETAILED DESCRIPTION:
The prevalence of diabetes is 7.4% in France among people aged 20 to 79 years in 2015. We must also consider "pre-diabetes" (subjects with glucose intolerance), whose prevalence is equivalent to that of diabetes (2012 estimate). The incidence of diabetes is exploding both for type 2 diabetes, which represents 85% of diabetes, and for type 1 diabetes, which represents 10% of cases and starts one out of two times before the age of 20. Diabetes typing is essential to guide therapeutic choices, particularly the use of insulin. This typing is based on the pathophysiology of the disease, distinguishing insulinopenia from autoimmune causes in type 1 diabetes, monogenic diabetes, secondary or atypical diabetes and type 2 diabetes, where insulinopenia and insulin resistance coexist. Thus, while a formal biological diagnosis is possible for some forms of atypical diabetes and for type 1 diabetes, no biological parameter is currently available for type 2 diabetes, which remains a diagnosis of exclusion. As a result, diabetes represents a source of diagnostic and therapeutic erraticism, amplified by the clinical heterogeneity of type 2 diabetes, which is obvious and underestimated, and by a clinical phenotyping of patients that is often defective. The economic consequences are important because the health costs are very different depending on whether or not patients are treated with insulin. Type 1 and type 2 diabetes are examples of chronic, non-transmissible, multigenic, multifactorial diseases. However, less than 10% of the heritability of type 2 diabetes is currently explained by the associated genetic variants. And although genetic tests exist to diagnose certain monogenic diabetes, this diagnosis is made in less than 20% of cases, mainly in the presence of an atypical clinical presentation of diabetes. Moreover, there is no reason to rule out the hypothesis of paucigenic forms, at the interface of monogenic diabetes and multigenic forms as usually envisaged, as has been observed in chronic pancreatitis, which is also accompanied by diabetes.

The study will be conducted according to a randomized trial design comparing two diagnostic strategies defined as follows:

* Control strategy: in silico analysis of a panel of validated genes (ISApanel - Diabetome 1). Patients recruited along the control procedure will stay in their group using current genetic diagnosis practices and standard of care that may differ from one center to another.
* Intervention strategy: whole genome sequencing coupled with multidisciplinary conciliation meeting.

We plan to randomize one patient in the control group for two in the intervention group.

The main objective of the study is to assess the contribution of whole genome sequencing (WGS) coupled with a multidisciplinary conciliation meeting (MCM) on diagnosis of atypical forms of diabetes compared to an in-silico analysis of a panel of validated genes (ISApanel), corresponding to current practice.

The target population is 1020 adults with atypical diabetes for whom it is possible to obtain a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years with confirmed diabetes mellitus according to WHO criteria (World Health Organization: Definition and diagnosis of diabetes mellitus and intermediate hyperglycemia: Report of a WHO/IDF Consultation. Geneva, World Health Org., 2006.)
* Age ≤ 45 years at diabetes diagnosis
* Body mass index ≤ 35 kg/m² at diabetes diagnosis
* Negative results of specific antibodies determination (GAD65, IA2, ZnT8) until the inclusion visit
* Presenting atypical diabetes defined by at least one of the following:
* Exocrine pancreatic disease
* Familial history: diabetes diagnosed in first degree relatives from at least 2 generations
* Notion of familial consanguinity
* Syndromic clinical features (dysmorphy, developmental delay, mental retardation…) or unusual abnormalities/features that are not part of diabetic complications or co-morbidities;
* Early occurrence of microvascular complications (≤ 5 years after diabetes diagnosis)
* Major insulinopenia at diagnosis (C peptide <0.2 nmol/L and/or documented ketosis)
* Patient who conserved endogenous insulin secretion (positive C peptide value) but a need for insulin therapy initiation during the first year following diagnosis due to therapeutic failure of well conducted therapeutic intensification
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Patient with a social security number in compliance with the French law (dispositions relatives aux recherches impliquant la personne humaine prévues aux articles L 1121-1 et suivants du Code de la Santé Publique)
* Signed and dated informed consent form

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Any contraindication to the study exams including known allergies or contraindication to contrasts for the scan
* Patient with known monogenic diabetes (defined as identification of class 4 and 5 variants according to ACMG)
* First or second-degree relatives with monogenic diabetes established by molecular genetics (class 4 and 5 variants according to ACMG)
* Patient with known secondary diabetes (i.e. endocrine disorders such as Cushing syndrome, pancreatectomy, drug-induced diabetes)
* Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol,
* Individuals under legal protection (sauvegarde de justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with one or several genetic alterations likely causal of diabetes | At 6 months in control group and 12 months in interventional group
  Number of patients in each group with one or several genetic alterations likely causal of diabetes

SECONDARY OUTCOMES:
Number of patients with an impact on treatment modification | 5 years
  Number of patients in each group with an impact on treatment modification including discontinuation and reason of this modification
Number of genetic alterations likely causal of diabetes | At 6 months in control group and 12 months in interventional group
  Number of genetic alterations likely causal of diabetes (classified as class 4 or 5 variants)
Feasibility of the whole genome sequencing (WGS) coupled with multidisciplinary conciliation meeting (MCM) on diagnosis of atypical forms of diabetes: time to access to the genetic data | At 6 months in control group and 12 months in interventional group
  time between blood sampling and availability of genetic data by GLUCOGEN laboratories
Feasibility of the WGS coupled with MCM on diagnosis of atypical forms of diabetes: time between blood sampling and MCM | At 6 months in control group and 12 months in interventional group
  time between blood sampling and MCM
Feasibility of the WGS coupled with MCM on diagnosis of atypical forms of diabetes: time between blood sampling and access to WGS report | At 6 months in control group and 12 months in interventional group
  time between blood sampling and access to WGS report produced by GLUCOGEN laboratory
Feasibility of the WGS coupled with MCM on diagnosis of atypical forms of diabetes: time between blood sampling and date of the WGS result visit | 5 years
  time between blood sampling and date of the WGS result visit
Genotype-Insulin secretion phenotype association | At 6 months in control group and 12 months in interventional group
  Genotype-phenotype associations corresponding to insulin secretion
Genotype-Insulin sensitivity phenotype association | At 6 months in control group and 12 months in interventional group
  Genotype-phenotype associations corresponding to insulin sensitivity
  • Body composition
Genotype-body composition phenotype association | At 6 months in control group and 12 months in interventional group
  Genotype-phenotype associations corresponding to body composition
Glycemic control without insulin treatment | 5 years
  Percentage of patients with glycated hemoglobin (HbA1c) target below 7% without insulin treatment at 2, 3, 4 and 5 years
Glycemic control without severe hypoglycemia | 5 years
  Percentage of patients with glycated hemoglobin (HbA1c) target below 7% without severe hypoglycemia in the last 6 months and with a change in body mass index < 1 kg/m² in the last 6 months at 2, 3, 4 and 5 years
Number of long-term micro and macro vascular complications associated with diabetes and time to occurrence of the first complication | 5 years
  Number of long-term micro and macro vascular complications associated with diabetes and time to occurrence of the first complication:
  * Retinopathy
  * Nephropathy
  * Neuropathy
  * Cardiovascular disease
  * Liver disease
Patient-Reported Outcomes (PROs), evaluated with SF36 questionnaire | 5 years
  SF36 questionnaire at baseline, every 6 months during the first 2 years, then every year until 5 years.
Patient-Reported Outcomes (PROs), evaluated with Euroquol Dimension (EQ-5D-5L) questionnaire | 5 years
  EQ-5D-5L questionnaire at baseline, every 6 months during the first 2 years, then every year until 5 years.
  • ADDQOL questionnaire
Patient-Reported Outcomes (PROs), evaluated with Audit of Diabetes Dependent Quality of Life (ADDQOL) questionnaire | 5 years
  ADDQOL questionnaire at baseline, every 6 months during the first 2 years, then every year until 5 years.
Number of participants agreeing to have access to secondary findings (SF) | At 6 months in control group and 12 months in interventional group
  Number of participants agreeing to have access to secondary findings (SF)
Number and type of SFs (class 4 or 5 variant(s)) identified in participants that specifically consent to have access to SF | At 6 months in control group and 12 months in interventional group
  Number and type of SFs (class 4 or 5 variant(s)) identified in participants that specifically consent to have access to SF
Percentage of SFs in the studied population | At 6 months in control group and 12 months in interventional group
  Percentage of SFs in the studied population
Number and type of medical consequences following identification of SFs | 5 years
  Number and type of medical consequences following identification of SFs
Direct costs associated with current diagnosis practices (ISApanel) | 5 years
  Direct costs associated with current diagnosis practices (ISApanel)
Direct costs associated with WGS coupled with MCM | 5 years
  Direct costs associated with WGS coupled with MCM
Incremental cost-effectiveness ratio of WGS coupled with MCM compared to current diagnosis practices (ISApanel) | 5 years
  Incremental cost-effectiveness ratio of WGS coupled with MCM compared to current diagnosis practices (ISApanel)
Incremental cost-utility ratio of WGS coupled with MCM compared to current diagnosis practices (ISApanel) | 5 years
  Incremental cost-utility ratio of WGS coupled with MCM compared to current diagnosis practices (ISApanel)
Cost-benefit of WGS coupled with MCM compared to current diagnosis practices | 5 years
  Cost-benefit of WGS coupled with MCM compared to current diagnosis practices (ISApanel) in terms of cost of wandering diagnosis and care procedure avoided
Psychosocial issues related to genetic testing for atypical diabetes | At 6 months in control group and 12 months in interventional group
  Qualitative data related to patients' expectations regarding genetic testing related to atypical diabetes and needs to receive SF information.
Psychosocial issues related to genetic testing for atypical diabetes | 5 years
  * Qualitative data (discourse - semi-structured individual interviews) related to patients experience following genetic testing results for atypical diabetes
  * Qualitative data (discourse - semi-structured individual interviews) related to patients' experience of the GLUCOGEN trial
Psychosocial issues related to patients' experience of the GLUCOGEN trial | 18 months
  Quantitative data (questionnaire)
Psychosocial issues related to professional's experience of the GLUCOGEN research protocol | 12 months
  Qualitative data (observation), including information regarding doctor-patient relationship and decision-making processes.

OTHER OUTCOMES:
Number and characteristics of new genomic variations responsible for diabetes development | At 6 months in control group and 12 months in interventional group
  Number and characteristics of new genomic variations responsible for diabetes development
Number and characteristics of genomic variations and their association with defined phenotypes including integrated diagnostic biomarkers | At 6 months in control group and 12 months in interventional group
  Number and characteristics of genomic variations and their association with defined phenotypes including integrated diagnostic biomarkers
Number and characteristics of genomic variations known as drug targets | At 6 months in control group and 12 months in interventional group
  Number and characteristics of genomic variations known as drug targets
Number and characteristics of genomic variations of metabolism, transport or drug targets of diabetes and their consequences on treatment response | At 6 months in control group and 12 months in interventional group
  Number and characteristics of genomic variations of metabolism, transport or drug targets of diabetes and their consequences on treatment response
Number and characteristics of molecular targets in atypical diabetes | At 6 months in control group and 12 months in interventional group
  Number and characteristics of molecular targets in atypical diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François GAUTIER, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (26):
- France (26):
  - University Hospital, Amiens
  - University Hospital, Angers
  - University Hospital Jean Minjoz, Besançon
  - University Hospital Haut Lévêque, Bordeaux
  - University Hospital Cavale Blanche, Brest
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - University Hospital Bocage, Dijon
  - University Hospital Michallon, Grenoble
  - Assistance Publique Hôpitaux de Paris, Bicêtre Hospital, Le Kremlin-Bicêtre
  - University Hospital Louis Pradel, Lyon
  - University Hospital Sud, Lyon
  - University Hospital Conception, Marseille
  - University Hospital Lapeyronie, Montpellier
  - University Hospital, Nancy
  - University Hospital Laennec, Nantes
  - University Hospital L'Archet, Nice
  - Assistance Publique Hôpitaux de Paris, Bichat - Claude Bernard Hospital, Paris
  - Assistance Publique Hôpitaux de Paris, Cochin Hospital, Paris
  - Assistance Publique Hôpitaux de Paris, Lariboisière Hospital, Paris
  - Assistance Publique Hôpitaux de Paris, Saint Antoine Hospital, Paris
  - Assistance Publique Hôpitaux de Paris- La Pitié Salpêtrière Hospital, Paris
  - University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - University Hospital Bois Guillaume, Rouen
  - Strasbourg University Hospital, Strasbourg
  - University Hospital Rangueil, Toulouse